CLINICAL TRIAL: NCT07189234
Title: TIMET 2.0 - Long Term Impact of Time-Restricted Eating on Parameters of Cardiometabolic Health
Brief Title: Long Term Impact of Time-Restricted Eating on Parameters of Cardiometabolic Health
Acronym: TIMET 2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 812281
Record Dates: First submitted 2025-09-04; First posted 2025-09-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome; Pre-diabetes
Keywords: Time Restricted Eating; Fasting
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Intermittent Fasting; Fasting | interventions — Trehalase; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (TRE) (Experimental): Participants in this arm will be asked to maintain their current lifestyle and medication management routines, while adhering to a daily, consistent 10-hour eating window. They will also receive standard lifestyle coaching, including meetings with a dietician to review dietary intake, and are required to track their caloric intake using a smartphone app.
  Interventions: Behavioral: Time-restricted eating (TRE) + Standard of Care
- Standard of care (SOC) (Placebo Comparator): Participants in this arm will maintain their current lifestyle and medication management without adhering to the 10-hour eating window. They will receive standard lifestyle coaching, including meetings with a dietician to review dietary intake, and will be asked to track their caloric intake using a smartphone app.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Time-restricted eating (TRE) + Standard of Care — Participants in this arm will adhere to a daily, consistent 10-hour eating window for the course of the study as well as receive nutritional counseling from the study dietician.
  Arms: Time-restricted eating (TRE)
Behavioral: Standard of Care — Participants in this arm will receive nutritional counseling from the study dietician, but will not be required to adopt the 10-hour eating window.
  Arms: Standard of care (SOC)

SUMMARY:
In a randomized controlled trial, the investigators intend to measure the health impact of time restricted eating (TRE) in patients with metabolic syndrome (with elevated blood pressure and at least 2 of the following: increased waist circumference, abnormal cholesterol levels, elevated triglycerides, and elevated fasting glucose levels), who habitually eat more than 12 hours every day. Patients will be randomly assigned to a control group (standard of care) or intervention group (TRE).

DETAILED DESCRIPTION:
Circadian rhythms optimize nutrient homeostasis by orchestrating catabolic and anabolic metabolism to appropriate times of the 24 hour day. Chronic circadian rhythm disruption predisposes individuals to metabolic diseases including obesity and type 2 diabetes. Conversely, maintaining a daily rhythm of feeding and fasting cycles sustains a robust circadian rhythm which improves cellular bioenergetics and results in improved metabolism. Time-restricted eating (TRE) is a specific feeding-fasting pattern in which feeding is restricted to 8-12 hours a day.

Over the 54-week duration of the study, participants will be required to use a smartphone application (myCircadianClock, developed by the Salk Institute) to log all food and beverage intake. Investigators will measure height, weight, waist circumference, and blood pressure throughout the study. Blood tests will be done after an overnight fast to check HbA1C, glucose, insulin, lipids, and an NMR lipoprotein profile. Blood sugar will also be monitored continuously using a continuous glucose monitor (CGM) worn for 2 weeks at the beginning of the study, at 6 months, and at 12 months (end of the study). At these same three timepoints, participants will also wear a wrist-worn actigraphy device (actiwatch) to track physical activity and sleep patterns. Body composition will be measured using a dual energy X-ray absorptiometry (DEXA) scan, and an oral glucose tolerance test (OGTT) will be performed to assess how the body responds to sugar.

ELIGIBILITY:
Inclusion criteria:

1. Age: 18-75 years
2. HbA1c: 5.7% to 7.0%
3. Metabolic syndrome (must meet 3 criteria):

   1. Elevated systolic blood pressure ≥ 130 mm Hg or diastolic blood pressure ≥ 85 mm Hg OR an antihypertensive therapy)
   2. Elevated waist circumference:

      - In Asians: ≥ 90 cm in men, ≥80 cm in women In all other races: ≥ 102 cm in men, ≥ 88 cm in women
   3. Fasting plasma triglycerides ≥ 150 mg/dL, or on drug treatment for elevated triglycerides d) Reduced High-density lipoprotein (HDL)- cholesterol < 40 mg/dL in males or < 50 mg//dL in females, or drug treatment for reduced HDL-cholesterol e) Fasting glucose ≥ 100 mg/dL
4. Own a smartphone (Apple iOS or Android OS)
5. Baseline eating period ≥12 hour/day
6. Patients on a stable dose of cardiovascular medications (HMG CoA reductase inhibitors [statins]), other lipid-modifying drugs (including over-the-counter drugs such as red yeast rice and fish oil), or anti-hypertensive drugs) for at least 1 month are allowed.
7. Patients on GLP-1 R agonists, SGLT2 inhibitors, or Metformin must be on stable doses for at least 3 months.

Exclusion criteria:

1. Use of sulfonylurea or insulin.
2. HbA1C > 7.0%
3. Pregnant or breastfeeding. Anyone of reproductive age will receive pregnancy test prior to DXA scan.
4. Caregiver for a dependent requiring frequent nocturnal care / sleep interruptions.
5. Shift workers with variable (e.g. nocturnal) hours.
6. Frequent travel to different time zones during the study period.
7. Active tobacco use or illicit drug use or history of treatment for alcohol abuse.
8. History of major adverse cardiovascular event within the past year (acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack).
9. History of surgical intervention for weight management within the past 2 years, or longer if deemed unsafe following review by medical investigators
10. Uncontrolled arrhythmia (i.e. rate -controlled atrial fibrillation / atrial flutter are not exclusion criteria)
11. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e. hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
12. History of adrenal disease.
13. History of malignancy undergoing active treatment, except non-melanoma skin cancer.
14. Known history of type 1 diabetes.
15. History of an eating disorder.
16. History of cirrhosis.
17. History of stage 4 or 5 chronic kidney disease or requiring dialysis.
18. Currently enrolled in a weight-loss or weight-management program.
19. On a special or prescribed diet for other reasons (e.g. Celiac disease).
20. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).
21. Inability or unwillingness to utilize the mCC app throughout study duration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2028-07-06 (Estimated); Study Completion 2029-01-06 (Estimated)

PRIMARY OUTCOMES:
Change in Glucose Levels | 54 weeks
  Assessed via HbA1c (%)

SECONDARY OUTCOMES:
Change in glycemic variability | 54 weeks
  Measured by continuous glucose monitor (CGM)
Change in direct LDL-C | 54 weeks
  LDL cholesterol (mg/dl)
Change in bone density | 54 weeks
  Bone density measured by DEXA scan (g/cm^2)
Change in insulin sensitivity | 54 weeks
  Measured by oral glucose tolerance test (OGTT)
Changes in muscle mass | 54 weeks
  Muscle mass measured by DEXA scan (kg)
Change in body fat | 54 weeks
  Measured by body fat percentage via DEXA scan (%)

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — UC San Diego Health
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

REFERENCES:
- [Background] Taub PR, Panda S. Time for better time-restricted eating trials to lessen the burden of metabolic diseases. Cell Rep Med. 2022 Jun 21;3(6):100665. doi: 10.1016/j.xcrm.2022.100665. PMID 35732151